CLINICAL TRIAL: NCT01757626
Title: Phase I/II Study of Combination Therapy of Antibody Hu3F8 With Granulocyte- Macrophage Colony Stimulating Factor (GM-CSF) in Patients With Relapsed/Refractory High-Risk Neuroblastoma
Brief Title: Combination Therapy of Antibody Hu3F8 With Granulocyte- Macrophage Colony Stimulating Factor (GM-CSF) in Patients With Relapsed/Refractory High-Risk Neuroblastoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-230
Record Dates: First submitted 2012-12-21; First posted 2012-12-31 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Neuroblastoma
Keywords: Bone Marrow; Hu3F8; GM-CSF; 12-230
MeSH Terms: conditions — Neuroblastoma | interventions — naxitamab; Granulocyte-Macrophage Colony-Stimulating Factor

ARMS (2):
- Hu3F8 with GM-CSF (Experimental): The phase I single arm trial assesses escalating doses of iv hu3F8 (days 1, 3, 5) in the presence of sc GM-CSF (day -4 through 5). These 3 doses of hu3F8 and 10 days of GM-CSF constitute a treatment cycle. The expansion phase II single arm trial assesses the anti-NB activity of hu3F8+GM-CSF.in 3 groups of patients: Group 1 patients have primary refractory disease (no prior relapse but incomplete response to treatment) in BM as documented by histology and/or 123I-MIBG scan. Group 2 patients are in ≥2nd CR and at high risk for another relapse. Group 3 patients have secondary refractory disease (prior relapse and incomplete response to retrieval therapy) in BM as documented by histology and/or 123I-MIBG scan. Ph II: Groups 1 & 3 pts can continue to get cycles every 1-2 months for up to 24 months from study enrollment or until they receive 5 cycles after a major response (CR or PR) is achieved.
  Interventions: Biological: Hu3F8 With GM-CSF
- expansion phase II single arm trial (Experimental): Group 1 patients have primary refractory disease (no prior relapse but incomplete response to treatment) in BM as documented by histology and/or 123^I-MIBG scan. Group 2 patients are in >2nd CR/VGPR and at high risk for another relapse. Group 3 patients have secondary refractory disease (prior relapse and incomplete response to retrieval therapy) in BM as documented by histology and/or 123^I-MIBG scan. GM-CSF can be omitted if patients have a history of an allergy to GM-CSF or develop an allergic reaction to GM-CSF after initiating therapy while on the protocol.
  Interventions: Biological: Hu3F8 With GM-CSF

INTERVENTIONS:
Biological: Hu3F8 With GM-CSF — Ph I: 1 cycle consists of treatment with hu3F8 for 3 days (day 1, 3 & 5). GM-CSF starts 5 days in advance of each hu3F8 cycle at 250 mcg/m^2/day (day -4 to day 0), & at 500 mcg/m^2/day x 5 days (day 1 to day 5). Hu3F8 cycles are 5 days. Ph II pts may receive treatment on a modified schedule of 3 doses of IV hu3F8 over a maximum of 10 days, as needed. With modified schedules of hu3F8, GM-CSF will be administered at 250 mcg/m2/day x5 days before the 1st dose of hu3F8, as with the standard schedule, but then GM-CSF at 500 mcg/m2/day will be administered on day of the 1st dose of hu3F8, on the day before and on the day of the 2nd dose of hu3F8, and on the day before and on the day of the 3rd dose of hu3F8. Cycles are repeated at 2-4 week intervals between 1st days of hu3F8, through 4 cycles. Pts who complete 4 cycles of treatment w/o complications or disease progression have the option of continuing treatment for up to 24 months from their 1st dose of hu3F8.
  Arms: Hu3F8 with GM-CSF
Biological: Hu3F8 With GM-CSF — As determined by the phase I component of the study, the hu3F8 dosage in the phase II portion is 3 mg/kg/day. Patients who were treated in the phase I component are eligible for treatment in the phase II portion. Cycles are repeated approximately monthly through 5 cycles. Group 1 and Group 3 patients can continue to receive cycles every 1-2 months for up to 24 months from study enrollment or until they receive 5 cycles after a major response (CR or PR) is achieved, whichever comes first. If HAHA becomes (+), cycles are deferred until it becomes (-) again. Patients who develop HAHA which precludes timely treatments with hu3F8+GM-CSF are eligible to receive low-dose maintenance regimens such as irinotecan alone,61 temozolomide alone,62 irinotecan-temozolomide,63 or cyclophosphamide-topotecan.64 They can also receive anti-HAHA agents such as rituximab and cyclophosphamide. They resume treatment with hu3F8+ GM-CSF if HAHA becomes negative. Patients may receive local radiation therapy.
  Arms: expansion phase II single arm trial

SUMMARY:
The purpose of this study is to find out if an antibody called Humanized 3F8 (Hu3F8) combined with granulocyte- macrophage colony stimulating factor (GM-CSF) is safe for treating neuroblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NB as defined by a) histopathology (confirmed by the MSKCC Department of Pathology), or b) BM metastases or MIBG-avid lesion(s) plus high urine catecholamine levels.
* Patients must have high-risk NB (including MYCNamplified stage 2/3/4/4S of any age and MYCN-nonamplified stage 4 in patients greater than 18 months of age) AND:
* Phase I: Patients must have refractory or relapsed NB, resistant to standard therapy*.

  *For NB, standard therapy includes intensive induction chemotherapy, followed by a variety of consolidation or salvage therapies, depending on response.
* Phase II: Patients must have primary or secondary refractory disease in BM, defined as morphologic evidence of NB in BM and/or abnormal 123I-MIBG uptake in osteomedullary sites, OR patients patients in ≥ 2nd CR patients are in ≥2nd CR
* Patients must be older than 1 year of age.
* Prior treatment with murine and humanized 3F8 is allowed. Patients with prior m3F8, hu3F8, ch14.18 or hu14.18 treatment must have a negative HAHA antibody titer. Human anti-mouse antibody (HAMA) positivity is allowed.
* White blood cell count ≥1000/ul (phase I only)
* Absolute neutrophil count ≥500/ul (phase I only)
* Absolute lymphocyte count ≥500/ul (phase I only)
* Platelet count ≥25,000/ul (phase I only)
* No chemotherapy or immunotherapy for a minimum of three weeks prior to start of hu3F8
* Women of child-bearing potential must be willing to practice an effective method of birth control while on treatment
* Signed informed consent indicating awareness of the investigational nature of this program.

Exclusion Criteria:

* Existing major organ dysfunction > grade 2, with the exception of hearing loss and hematologic toxicity (defined as suppression of all subtypes of WBCs, RBCs, and platelets).
* Active life-threatening infection.
* Pregnant women or women who are breast-feeding.
* Inability to comply with protocol requirements, including PK studies and genetic studies (phase I only)
* History of allergy to mouse proteins.
* Positive human anti-hu3F8 antibody (HAHA) titer

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2012-12; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dosage | 1 year
  hu3F8 when combined with GM-CSF. DLT is defined after 1 cycle. Seventeen dosage levels of hu3F8 will be tested with three to six patients at each dosage level.
assess the toxicity | 1 year
  of the humanized anti GD2 antibody hu3F8 when combined with Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) in patients with high risk neuroblastoma. All observed adverse events, regardless of treatment group or suspected causal relationship to study drug will be recorded. Adverse events will be identified and graded using the Common Toxicity Criteria Version 4.0

SECONDARY OUTCOMES:
pharmacokinetics of hu3F8 | 1 year
  (Phase I) when combined with GM-CSF. Pharmacokinetics will be measured by serial blood sampling following the first two iv doses of hu3F8 as listed in Table 3. Serum hu3F8 will be measured pre-infusion and at time pre- (within an hour before hu3F8), 5 min, 3h, 6-8h, 24h, 48h, 72h, 96, 120h, 168h 216h and 264h after the first infusion of hu3F8 during cycle1 and, whenever possible, peak hu3F8 level at pre- and ~5 minutes post-infusion will also be measured for each dose of hu3F8 in subsequent cycles .
assess activity of hu3F8 plus GM-CSF against HR-NB | 2 years
  Another secondary objective is to assess the anti-tumor activity of hu3F8 against NB and other GD2-positive tumors. Anti-tumor activity will be measured by international neuroblastoma response criteria (INRC).
quantitate the response of marrow NB | 1 year
  will be measured using quantitative Reverse transcription-PCR (qRTPCR) and its relationship with dosage of hu3F8 explored.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kushner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Kushner BH, Modak S, White C, Basu EM, Roberts SS, Mauguen A, Cheung NV. A phase II trial of naxitamab plus stepped-up dosing of GM-CSF for patients with high-risk neuroblastoma in second or later complete remission. Int J Cancer. 2026 Feb 11. doi: 10.1002/ijc.70374. Online ahead of print. PMID 41670398
- [Derived] Kushner BH, Modak S, Mauguen A, Basu EM, Roberts SS, Cheung NV. Naxitamab plus stepped-up dosing of granulocyte-macrophage colony-stimulating factor for primary refractory high-risk neuroblastoma: results of a phase I/II trial. J Hematol Oncol. 2025 Nov 26;18(1):114. doi: 10.1186/s13045-025-01770-7. PMID 41299684
- [Derived] Kushner BH, Cheung IY, Modak S, Basu EM, Roberts SS, Cheung NK. Humanized 3F8 Anti-GD2 Monoclonal Antibody Dosing With Granulocyte-Macrophage Colony-Stimulating Factor in Patients With Resistant Neuroblastoma: A Phase 1 Clinical Trial. JAMA Oncol. 2018 Dec 1;4(12):1729-1735. doi: 10.1001/jamaoncol.2018.4005. PMID 30326045
- [Derived] Cheung IY, Kushner BH, Modak S, Basu EM, Roberts SS, Cheung NV. Phase I trial of anti-GD2 monoclonal antibody hu3F8 plus GM-CSF: Impact of body weight, immunogenicity and anti-GD2 response on pharmacokinetics and survival. Oncoimmunology. 2017 Jul 31;6(11):e1358331. doi: 10.1080/2162402X.2017.1358331. eCollection 2017. PMID 29147617
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/